CLINICAL TRIAL: NCT04142515
Title: Collection and Analysis of the Clinical and Biological Characteristics of Patients Treated at Nîmes Carémeau University Hospital, for Giant Cells ARTEitis (Horton's Disease), for Diagnosis and During Long-term Follow-up
Brief Title: Collection and Analysis of the Clinical and Biological Characteristics of Patients Treated for Giant Cells ARTEitis (Horton's Disease)
Acronym: CARTECEL
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: Local2019/RG-01
Record Dates: First submitted 2019-10-25; First posted 2019-10-29 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Giant Cell Arteritis; Horton Disease
MeSH Terms: conditions — Giant Cell Arteritis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Giant cell arteritis (GCA) or Horton's disease: frequent large vessel vasculitis (cephalic) (incidence estimated at 9 per 100,000 in France), potentially responsible for blindness.

Treatment: corticosteroid therapy, which is effective in the vast majority of cases.

Clinical problem: relapse; 36% to 44% of patients have a relapse that occurs in the first year for many patients, requiring a re-escalation of corticosteroid therapy, with its consequences:

* Cumulative dose of corticosteroid therapy that causes cardiovascular and infectious morbidity.
* Requires additional immunosuppressive treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 45 years or older
* Patients with giant cell arteritis according to ACR criteria or revised criteria incorporating imaging parameters,
* Patients managed at the University Hospital of Carémeau in Internal Medicine from 01/01/2011 to 01/01/2020.

Exclusion Criteria:

None

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 45 years or older with giant cell arteritis according to ACR criteria or revised criteria incorporating imaging parameters, managed at the University Hospital of Carémeau in Internal Medicine from 01/01/2011 to 01/01/2020.
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Clinical and paraclinical characteristics of patients diagnosed with ACG | day 1
  Describe the clinical and paraclinical characteristics of patients diagnosed with ACG to determine whether certain characteristics are significantly associated with a higher risk of developing corticosteroid dependence

CONTACTS AND LOCATIONS:
Locations (1):
- CHUNimes, Nîmes, France

IPD SHARING:
Plan to Share IPD: Undecided